CLINICAL TRIAL: NCT06056024
Title: Open-label Dose-finding Trial to Explore Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of BI 3706674 Given Orally as Monotherapy in Patients With Unresectable Metastatic KRAS Wild Type Amplified Gastric, Oesophageal, and Gastroesophagealjunction Adenocarcinoma
Brief Title: A Study to Test How Well Different Doses of BI 3706674 Are Tolerated by People With Advanced Cancer in the Stomach and Oesophagus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1512-0001
Record Dates: First submitted 2023-09-19; First posted 2023-09-28 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumor, KRAS Mutation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A (Phase Ia): Dose escalation (Experimental)
  Interventions: Drug: BI 3706674
- Part B (Phase Ib): Dose confirmation (Experimental)
  Interventions: Drug: BI 3706674
- Part C (Phase Ib): Dose expansion (Experimental)
  Interventions: Drug: BI 3706674

INTERVENTIONS:
Drug: BI 3706674 — BI 3706674

SUMMARY:
This study is no longer open to new participants. It was a study in adults with advanced cancer in the stomach and oesophagus. This is a study for people for whom previous treatment was not successful or no treatment exists. In this study, BI 3706674 is given to humans for the first time.

The purpose of this study is to find a suitable dose of BI 3706674 that people with advanced cancer can tolerate when taken alone. Another purpose is to check whether BI 3706674 can make tumours shrink. BI 3706674 blocks growth signals and may prevent the tumour from growing.

Participants take BI 3706674 as a tablet when starting treatment. Different doses of BI 3706674 are tested during this study. If there is benefit for the participants and if they can tolerate it, the treatment is given up to the maximum duration of the study. During this time, participants visit the study site regularly. The total number of visits depends on how they respond to and tolerate the treatment. Doctors record any unwanted effects and regularly check the general health of the participants.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologically confirmed diagnosis of locally advanced or metastatic gastric adenocarcinoma (GAC), oesophageal adenocarcinomas (EAC), and gastroesophageal junction adenocarcinoma (GEJAC) with Kirsten rat sarcoma viral oncogene homolog (KRAS) wild type (wt) amplification and documented disease progression despite at least 1 line of prior therapy. KRAS status will be confirmed retrospectively for those with a known KRAS status or determined prospectively (dose confirmation and expansion) if KRAS status is unknown, using archival tissue (if available) or a fresh biopsy.

   Dose escalation (Part A) only: Patients with advanced or metastatic relapsed or refractory solid tumours of any histology with KRAS wt amplification or harbouring a KRAS G12V mutation who have exhausted treatment options known to prolong survival for their disease. Detection of KRAS status by a local test is allowed for enrolment but will be retrospectively confirmed.
2. Patients who have failed conventional treatment or for whom no therapy of proven efficacy exists or who are not eligible for established treatment options.
3. Dose confirmation (Part B) only: Patient is willing and able to undergo mandatory pre- and on-treatment low risk tumour biopsies. Patients with a high risk for biopsy complications can be included without undergoing pre- and on-treatment tumour biopsy as long as archival tumour tissue is available for confirmation of KRAS status.
4. At least one target lesion that can be measured per RECIST version 1.1 (radiated lesions do not qualify as target lesions unless there has been demonstrated progression of the lesion after completion of radiotherapy) Dose escalation (Part A) only: Patients with no lesions measurable per RECIST version 1.1 may be included if agreed between Sponsor and investigator.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. All toxicities related to previous anti-cancer therapies have resolved ≤ CTCAE Grade 1 prior to trial treatment administration (except for alopecia and peripheral neuropathy which must be ≤ CTCAE Grade 2 and amenorrhea/menstrual disorders which can be any grade).
7. Life expectancy ≥3 months at the start of treatment in the opinion of the investigator.
8. Age ≥18 years of age, or over the legal age of consent as required by local legislation.

Further inclusion criteria apply.

Exclusion Criteria:

1. Previous anti-cancer chemotherapy within 3 weeks of the first administration of trial drug.
2. Previous anti-cancer hormonal treatment or anti-cancer immunotherapy within 2 weeks of the first administration of trial drug.
3. Previous treatment with rat sarcoma (RAS), mitogen-activated protein kinases (MAPKs) or son of sevenless homolog 1 (SOS1) targeting agents.
4. Presence of cardiovascular abnormalities such as uncontrolled hypertension (defined as systolic blood pressure ≥140 and/or diastolic blood pressure ≥90 millimetre of mercury (mmHg)), congestive heart failure New York Heart Association (NYHA) classification of ≥ III or IV, unstable angina or poorly controlled arrhythmia. History of myocardial infarction, stroke, or pulmonary embolism within 6 months prior to randomisation.
5. Left ventricular ejection fraction (LVEF) <50%.
6. Congenital or family history of long QT prolongation syndrome.
7. Mean resting corrected QT interval (QTcF) >470 msec.
8. Radiotherapy within 2 weeks prior to start of treatment, except as follows:

   * Palliative radiotherapy to regions other than the chest is allowed if completed at least 2 weeks prior to randomisation.
   * Single dose palliative radiotherapy for symptomatic metastasis within 2 weeks prior to randomisation may be allowed but must be discussed with the Sponsor.

Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-12-06 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
Part A: Occurrence of dose limiting toxicities (DLTs) in the maximum tolerated dose (MTD) evaluation period | up to 28 days
Part B: Occurrence of drug-related adverse events (AEs) ≥ Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 during the on-treatment period | up to 3.5 years
Part C: Objective response (OR) based on central assessment | up to 3.5 years
  OR is defined as best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR), where BOR is determined according to Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1 from first treatment administration until the earliest of disease progression, death, or last evaluable tumour assessment before start of subsequent anticancer therapy, loss to follow-up or withdrawal of consent.

SECONDARY OUTCOMES:
Part A: Occurrence of DLTs during the on-treatment period | up to 3.5 years
Part B: Occurrence of DLTs during the on-treatment period | up to 3.5 years
Part B: OR based on central assessment | up to 3.5 years
  OR is defined as best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR), where BOR is determined according to Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1 from first treatment administration until the earliest of disease progression, death, or last evaluable tumour assessment before start of subsequent anticancer therapy, loss to follow-up or withdrawal of consent.
Part B: Duration of objective response (DOR) | up to 3.5 years
  DOR is defined as the time from first documented CR or PR until the earliest of disease progression or death among patients with objective response.
Part B: Tumour shrinkage | up to 3.5 years
  Tumour shrinkage is defined as the difference between the minimum post-baseline sum of diameters of target lesions (long axis for non-nodal lesions, short axis for nodal lesions) and the baseline sum of diameters of the same set of target lesions.
Part B: Progression-free survival (PFS) | up to 3.5 years
  PFS is defined as the time from first treatment administration until tumour progression according to RECIST version 1.1 or death from any cause, whichever occurs earlier.
Part C: Duration of objective response | up to 3.5 years
Part C: Tumour shrinkage | up to 3.5 years
Part C: Progression-free survival (PFS) | up to 3.5 years
All trial parts: Maximum measured concentration (Cmax) of BI 3706674 evaluated after the first dose in Cycle 1 | up to 28 days
All trial parts: Area under the plasma concentration-time curve over a uniform dosing interval τ (AUCτ) of BI 3706674 evaluated after the first dose in Cycle 1 | up to 28 days
Maximum measured concentration of BI 3706674 evaluated at steady state on Cycle 2 Day 1 (Cmax,ss) | From Day 1 of Cycle 2 (each cycle is 28 days) up to 3.5 years
All trial parts: Area under the plasma concentration-time curve over a uniform dosing interval τ of BI 3706674 evaluated at steady state on Cycle 2 Day 1 (AUCτ,ss) | From Day 1 of Cycle 2 (each cycle is 28 days) up to 3.5 years
All trial parts: Occurrence of AEs during the on-treatment period | up to 3.5 years

CONTACTS AND LOCATIONS:
Locations (17):
- United States (6):
  - Mayo Clinic-Arizona, Phoenix, Arizona
  - Yale Cancer Center, New Haven, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Japan (2):
  - National Cancer Center Hospital East, Chiba, Kashiwa
  - Japanese Foundation for Cancer Research, Tokyo, Koto-ku
- South Korea (7):
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul
  - Ajou University Hospital, Suwon
- Taiwan (2):
  - NCKUH, Tainan
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.clinicalstudies.boehringer-ingelheim.com/msw/datatransparency